CLINICAL TRIAL: NCT06876714
Title: ShortStop-HER2: Shortened Duration of Adjuvant Therapy in Patients With Early-Stage HER2+ Breast Cancer Who Achieve pCR After Neoadjuvant Chemotherapy With HER2 Blockade
Brief Title: ShortStop-HER2: 12 Months vs. 6 Months of HER2-targeted Medications for People With HER2+ Breast Cancer Who Had a Pathologic Complete Response After Chemotherapy Plus Trastuzumab
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A012303; NCI-2024-10478 (Other: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Early Stage Breast Carcinoma
MeSH Terms: interventions — Trastuzumab; pertuzumab; High-Energy Shock Waves; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (12-month adjuvant therapy) (Active Comparator): Patients receive trastuzumab IV or SC on day 1 of each cycle. Patients may also receive pertuzumab IV or SC, at the discretion of the treating investigator, on day 1 of each cycle. Cycles repeat every 21 days for up to 17 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo ECHO or MUGA as well as mammography, ultrasound, or MRI throughout the trial. Patients may also optionally undergo blood and tissue sample collection throughout the trial.
  Interventions: Biological: Trastuzumab (Herceptin); Biological: Pertuzumab; Procedure: Echocardiography; Procedure: Multigated Acquisition Scan; Procedure: Mammography; Procedure: Ultrasound; Procedure: Magnetic Resonance Imaging; Procedure: Biospecimen Collection; Other: Questionnaire Administration
- Arm 2 (6-month adjuvant therapy) (Experimental): Patients receive trastuzumab IV or SC on day 1 of each cycle. Patients may also receive pertuzumab IV or SC, at the discretion of the treating investigator, on day 1 of each cycle. Cycles repeat every 21 days for up to 9 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo ECHO or MUGA as well as mammography, ultrasound, or MRI throughout the trial. Patients may also optionally undergo blood and tissue sample collection throughout the trial.
  Interventions: Biological: Trastuzumab (Herceptin); Biological: Pertuzumab; Procedure: Echocardiography; Procedure: Multigated Acquisition Scan; Procedure: Mammography; Procedure: Ultrasound; Procedure: Magnetic Resonance Imaging; Procedure: Biospecimen Collection; Other: Questionnaire Administration

INTERVENTIONS:
Biological: Trastuzumab (Herceptin) — Given IV or SC
Biological: Pertuzumab — Given IV or SC
Procedure: Echocardiography — Undergo ECHO
Procedure: Multigated Acquisition Scan — Undergo MUGA
Procedure: Mammography — Undergo mammography
Procedure: Ultrasound — Undergo ultrasound
Procedure: Magnetic Resonance Imaging — Undergo MRI
Procedure: Biospecimen Collection — Undergo blood and tissue sample collection
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial compares 6 months of human epidermal growth factor receptor 2 (HER2)-targeted therapy to 12 months of HER2-targeted therapy for the treatment of HER2-positive (+) breast cancer in patients that had a pathologic complete response (pCR) after preoperative (neoadjuvant) chemotherapy with trastuzumab. Trastuzumab and pertuzumab are monoclonal antibodies and forms of targeted therapy that attach to a receptor protein called HER2. HER2 is found on some cancer cells. When trastuzumab or pertuzumab attach to HER2, the signals that tell the cells to grow are blocked and the tumor cell may be marked for destruction by the body's immune system. Giving 6 months of HER2-targeted therapy may work better than giving 12 months for the treatment of HER2+ breast cancer in patients that had a pCR after neoadjuvant chemotherapy with trastuzumab.

DETAILED DESCRIPTION:
The primary and secondary objectives of the study:

PRIMARY OBJECTIVES:

I. To evaluate whether 6 months of combined neoadjuvant (neo)/adjuvant HER2 blockade results in a non-inferior recurrence-free survival (RFS) compared to 12 months of combined neo/adjuvant HER2 blockade, in patients with early stage HER2+ breast cancer who achieve pCR after neoadjuvant chemotherapy with HER2 blockade.

II. To compare the Functional Assessment of Cancer Therapy-Breast (FACT-B) total score at 12 months between patients randomized to receive 6 months versus 12 months of combined neo/adjuvant HER2 blockade. (Quality of life)

SECONDARY OBJECTIVES:

I. Secondary objectives are to evaluate whether 6 months compared to 12 months results in differences for the following:

Ia. Grade 3 or higher adverse event (AE) rates; Ib. Overall survival (OS); Ic. Locoregional recurrence (LRR, both isolated LRR as first events, and LRR events simultaneous with distant metastasis [DM]) incidence; Id. RFS for key subgroups: baseline stage, hormone receptor (HR) status, neoadjuvant chemotherapy backbone, and dual versus single HER2 blockade in the adjuvant setting; Ie. Time to central nervous system (CNS) recurrence (both isolated CNS recurrence as first events, and CNS recurrence events simultaneous with distant metastasis and/or LRR).

II. To compare the FACT-B total score at 18 months between patients randomized to receive 6 months versus 12 months of combined neo/adjuvant HER2 blockade. (Quality of life) III. To compare side effect bother as measured by the Functional Assessment of Cancer Therapy General Population 5 (FACT GP5) item at 12 months between patients randomized to receive 6 months versus 12 months of combined neo/adjuvant HER2 blockade. (Quality of life) IV. To compare specific patient-reported symptomatic adverse events (i.e. diarrhea, constipation, fatigue, and rash) as measured by the Patient Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) at 12 months between patients randomized to receive 6 months versus 12 months of combined neo/adjuvant HER2 blockade. (Quality of life)

QUALITY OF LIFE EXPLORATORY OBJECTIVES:

I. To examine the different FACT-B subscales at all other evaluable time points.

II. To examine heterogeneity of treatment effects within subgroups defined by subcutaneous versus intravenous treatment delivery.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive trastuzumab intravenously (IV) or subcutaneously (SC) on day 1 of each cycle. Patients may also receive pertuzumab IV or SC, at the discretion of the treating investigator, on day 1 of each cycle. Cycles repeat every 21 days for up to 17 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo echocardiography (ECHO) or multigated acquisition (MUGA) as well as mammography, ultrasound, or magnetic resonance imaging (MRI) throughout the trial. Patients may also optionally undergo blood and tissue sample collection throughout the trial.

ARM 2: Patients receive trastuzumab IV or SC on day 1 of each cycle. Patients may also receive pertuzumab IV or SC, at the discretion of the treating investigator, on day 1 of each cycle. Cycles repeat every 21 days for up to 9 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo ECHO or MUGA as well as mammography, ultrasound, or MRI throughout the trial. Patients may also optionally undergo blood and tissue sample collection throughout the trial.

After completion of study treatment, patients are followed up every 6 months for 5 years after registration or until recurrence and then annually for a total of 10 years after registration.

ELIGIBILITY:
Inclusion Criteria:

* Patients (females and males) with clinical stage T1c-T3 (or Tx) and nodal stage N0-N1 (except T3N1 tumors, which are not eligible)
* Patients must have no residual invasive disease in the breast or lymph nodes after the completion of neoadjuvant therapy. Residual ductal carcinoma in situ (DCIS) is allowed. Patients with residual isolated tumor cells at surgery are considered node-positive and are not eligible
* HER2+ by American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines. Central pathology review is not required. In cases where there were multiple tumor sites in breast/nodes that had HER2 testing at diagnosis, at least one site must have been HER2+ AND the treating investigator must feel it is in the patient's best interest to be treated as having HER2+ breast cancer
* Known hormone receptor status as defined by ASCO/CAP guidelines. Estrogen receptor (ER) and progesterone receptor (PR) of any values are allowed. Hormone receptor positive status can be determined by either known positive ER or known positive PR status; hormone receptor negative status must be determined by both known negative ER and known negative PR
* If invasive disease was present in both breasts, participation in the study is permitted as long as the eligibility criteria are met for both tumors/breasts (including the requirement that at least one biopsied site on each side must have been HER2+)
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patients must have received neoadjuvant chemotherapy in combination with trastuzumab with or without pertuzumab for a minimum of 12 weeks. All chemotherapy must have been completed preoperatively

  * Patient must complete a minimum of 12 weeks of coverage with trastuzumab and a maximum of 24 weeks in the combined neoadjuvant and adjuvant setting prior to trial registration. Trastuzumab may have been administered either weekly or once every 3 weeks (q3weeks). (For purposes of this eligibility criterion, a single dose of q3week trastuzumab would provide 3 weeks of coverage; a single dose of once a week (q1week) trastuzumab would provide 1 week of coverage. If a q3week dose of trastuzumab were administered and then the subsequent dose was delayed for any period of time, that would still count as 3 weeks of coverage.)
  * Administration of endocrine therapy for treatment of this breast cancer is allowed prior to trial registration. If a patient received prior breast cancer endocrine therapy (eg tamoxifen or aromatase inhibitor) for DCIS or preventive indication, and endocrine therapy is indicated for treatment of their current breast cancer, then prior endocrine therapy must have been stopped > 12 months prior to registration on this protocol
  * No use of investigational anti-cancer agents at time of registration
* Patient must register within 14 weeks of final surgery
* Adequate excision: Surgical removal of all clinically evident disease in the breast and lymph nodes as follows:

  * Breast surgery: Total mastectomy with grossly negative margins (in the opinion of the surgeon there is no disease grossly at the margins) or breast-conserving surgery with histologically negative margins (no ink on tumor, including DCIS) unless those margins are anterior at the skin or posterior at the chest wall and no additional margin re-excision can be performed
  * Lymph node surgery: Lymph node surgery must have been performed and can include sentinel lymph node biopsy, targeted axillary dissection, or axillary dissection, at the discretion of the breast surgeon
* Adequate radiation: Patients who completed breast-conserving surgery (i.e. lumpectomy) must have received or plan to receive adjuvant radiation. If breast-conserving surgery was performed but patient will not be receiving breast radiation, the patient is not eligible. Patients for whom radiotherapy would be recommended for breast cancer treatment but for whom it is contraindicated because of medical reasons (e.g., connective tissue disorder or prior ipsilateral breast radiation) are not eligible

  * Adjuvant radiation can be given on study, and in this case is encouraged to be given concurrently with adjuvant HER2-directed therapy, per investigator discretion
  * Targeting of the regional nodal basins will be at treating investigator discretion
* Not pregnant and not nursing, because this study involves agents with known teratogenic potential. Therefore, for women of childbearing potential only, a negative serum or urine pregnancy test should be performed prior to receiving HER2-directed therapy according to local standard practice
* Adequate hepatic, renal and bone marrow function to receive adjuvant HER2-directed therapy in the opinion of the treating investigator. There are no specific required laboratory values for eligibility
* No stage IV (metastatic) breast cancer
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* No history of any prior (ipsilateral [ipsi-] or contralateral) invasive breast cancer. Prior DCIS is allowed
* No evidence of recurrent disease following preoperative therapy and surgery
* Patients living with HIV who are healthy and deemed by their medical team to have a low risk of AIDS-related illnesses are included in this trial. Patients with Hepatitis B or Hepatitis C virus who are healthy and deemed by their medical team to meet all other enrollment criteria are included in this trial.
* Patients with inadequate cardiac function on most recent assessment of left ventricular ejection fraction (LVEF) are not eligible for this trial. Inadequate cardiac function is defined as LVEF < 50% on echocardiogram (echo) or multiple-gated acquisition (MUGA)
* No history of grade 3 or 4 toxicity related to trastuzumab. If pertuzumab is planned to be given on trial, patient must also have no history of grade 3-4 toxicity related to pertuzumab
* No contraindication to receipt of further HER2-directed therapy
* No patients with severe, uncontrolled systemic disease that may interfere with planned trial therapy.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1524 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2028-03-13 (Estimated); Study Completion 2037-03-13 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival (RFS) | From randomization to invasive local, regional or distant breast cancer recurrence, or death from any cause prior to a documented disease recurrence, assessed up to 10 years
  The Kaplan-Meier method will be used to estimate the distribution of RFS times and a stratified log-rank test for non-inferiority will be used to assess whether RFS with 6 total months of human epidermal growth factor receptor 2 (HER2)-blockade is non-inferior to standard-of-care 12 total months of HER2-blockade in this patient population. Stratified Cox modeling will be used to estimate the hazard ratio and corresponding one-sided 95% confidence interval (CI).
Functional Assessment of Cancer Therapy-Breast (FACT-B) total score (Quality of life) | At 12 months
  Will compare the FACT-B total score between patients randomized to receive 6 months versus 12 months of combined neoadjuvant/adjuvant HER2 blockade. All questionnaires will be scored according to published scoring algorithms, including recommendations for addressing missing items within a scale. An intention-to-treat (ITT) approach will be used for all analyses. All statistical tests will be 2-sided, and p-values < 0.05 will be considered statistically significant. To evaluate the between-arm mean difference in scores, a repeated measures mixed model will be estimated based on FACT-B total scores at all time points.

SECONDARY OUTCOMES:
Incidence of grade 3 or higher adverse events (AE) | Baseline to 30 days after last dose of study treatment
  Will be according to the Common Terminology Criteria for Adverse Events version 5.0. The maximum grade of a specific AE experienced by a patient will be used. The proportion of patients who report a grade 3 or higher AE will be compared between the two treatment arms with a chi-square test. AEs (type and grade) for both arms will be summarized with the frequency and relative frequency
Locoregional recurrence (LRR) | From randomization until invasive tumor recurs in the ipsilateral breast or chest wall, axillary, supraclavicular, or internal mammary nodes (if before or synchronous with a systemic recurrence), whichever comes first, assessed up to 10 years
  The cumulative incidence of LRR will be analyzed with Kaplan-Meier estimates (curve starting at 0 rather than 1) and compared with a stratified log rank test.
Overall survival | From randomization until death due to any cause, assessed up to 10 years
  Will be compared between the treatment arms with a stratified log rank test and a stratified Cox model will be used to generate the hazard ratio estimate (both a point estimate and 95% CI). The analyses will be done as ITT groups as well as per-protocol groups.
RFS for key subgroups | From randomization to invasive local, regional or distant breast cancer recurrence, or death from any cause prior to a documented disease recurrence, assessed up to 10 years
  Forest plots will be generated for key prognostic variables (including the stratification variables) and subgroups of interest to determine whether the treatment effect appears homogeneous across the subgroups for the ITT population. Additional key subgroups of interest are neoadjuvant chemotherapy backbone and the type of adjuvant HER2-blockade the patient actually received (dual versus single). With respect to the latter analysis, the interest will be in whether there is an apparent difference in treatment effect among patients who received adjuvant pertuzumab versus those who did not.
Time to central nervous system (CNS) recurrence | up to 10 years
  Will assess both isolated CNS recurrence as first events, and CNS recurrence events simultaneous with distant metastasis and/or LRR.
FACT-B total score (Quality of life) | At 18 months
  Will compare the FACT-B total score between patients randomized to receive 6 months versus 12 months of combined neo/adjuvant HER2 blockade. All questionnaires will be scored according to published scoring algorithms, including recommendations for addressing missing items within a scale. An ITT approach will be used for all analyses. All statistical tests will be 2-sided, and p-values <0.05 will be considered statistically significant. To evaluate the between-arm mean difference in scores, a repeated measures mixed model will be estimated based on FACT-B total scores at all time points.
Side effect bother (Quality of life) | At 6 or 12 months
  Will be assessed by Functional Assessment of Cancer Therapy General Population 5 between patients randomized to receive 6 months versus 12 months of combined neo/adjuvant HER2 blockade. All questionnaires will be scored according to published scoring algorithms, including recommendations for addressing missing items within a scale. An ITT approach will be used for all analyses. All statistical tests will be 2-sided, and p-values <0.05 will be considered statistically significant. To evaluate the between-arm mean difference in scores, a repeated measures mixed model will be estimated based on scores. Mean trajectories over time will be plotted by arm.
Patient reported symptomatic AE (Quality of life) | At 6 or 12 months
  Will be measured by Patient Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE). Will assess symptomatic AE using PRO-CTCAE measures for symptoms of interest, specifically diarrhea, constipation, fatigue, and rash. The proportion of patients with a maximum post-baseline score greater than 0 will be compared between arms using Fisher's exact test. For diarrhea, constipation, and fatigue, the proportion of patients with a maximum post-baseline score greater than or equal to 3 will be compared between arms using Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne Waks, MD, Study Chair — Alliance for Clinical Trials in Oncology
Locations (487):
- United States (483):
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Enloe Medical Center, Chico, California
  - Kaiser Permanente Dublin, Dublin, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Mercy Cancer Center, Merced, California
  - Kaiser Permanente- Modesto MOB II, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Joseph's Medical Center, Stockton, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - UCI Health - Yorba Linda, Yorba Linda, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Shaw Cancer Center, Edwards, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Saint Anthony North Hospital, Westminster, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - The Watson Clinic, Lakeland, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - South Florida Baptist Hospital, Plant City, Florida
  - Saint Anthony's Hospital Cancer Care Center, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Winter Haven Hospital, Winter Haven, Florida
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - UChicago Medicine AdventHealth Cancer Institute Hinsdale, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Trinity Medical Center, Moline, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - IU Health West Hospital, Avon, Indiana
  - IU Health North Hospital, Carmel, Indiana
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - UI Healthcare Mission Cancer and Blood - Pella, Pella, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - The Iowa Clinic PC, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Saint Joseph Mount Sterling, Mount Sterling, Kentucky
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - MaineHealth Cancer Care and IV Therapy - Brunswick, Brunswick, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - UM Upper Chesapeake Hematology and Oncology - Aberdeen, Aberdeen, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - MedStar Health Bel Air Medical Campus, Bel Air, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - MedStar Southern Maryland Hospital Center, Clinton, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - MedStar Montgomery Medical Center, Olney, Maryland
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - Briarcliff, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Hi-Line Sletten Cancer Center, Havre, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Jefferson Cherry Hill Hospital, Cherry Hill, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Novant Health Colon and Rectal Clinic, Clemmons, North Carolina
  - Novant Health Breast Surgery - Greensboro, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Novant Health Cancer Institute - Huntersville, Huntersville, North Carolina
  - Novant Health Presbyterian Medical Center Huntersville, Huntersville, North Carolina
  - Novant Health Cancer Institute - Kernersville, Kernersville, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Institute - Matthews, Matthews, North Carolina
  - Novant Health Cancer Institute - Mooresville, Mooresville, North Carolina
  - Novant Health Cancer Institute - Mount Airy, Mount Airy, North Carolina
  - Novant Health Cancer Institute - Wilkesboro, North Wilkesboro, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Novant Health Cancer Institute - Rowan, Salisbury, North Carolina
  - Rowan Regional Medical Center, Salisbury, North Carolina
  - Novant Health Cancer Institute - Statesville, Statesville, North Carolina
  - Novant Health Cancer Institute - Thomasville, Thomasville, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Aultman Alliance Community Hospital, Alliance, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Hood River Memorial Hospital, Hood River, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - UPMC Hillman Cancer Center at Butler Health System, Butler, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Chambersburg, Pennsylvania
  - UPMC Hillman Cancer Center - Passavant - Cranberry, Cranberry Township, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - IRMC Cancer Center, Indiana, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - Arnold Palmer Cancer Center Medical Oncology Norwin, N. Huntingdon, Pennsylvania
  - UPMC Hillman Cancer Center - New Castle, New Castle, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Cancer Center-Uniontown, Uniontown, Pennsylvania
  - UPMC Cancer Center-Washington, Washington, Pennsylvania
  - UPMC West Mifflin-Cancer Center Jefferson, West Mifflin, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Divine Providence Hospital, Williamsport, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Houston Methodist San Jacinto Hospital, Baytown, Texas
  - MD Anderson in The Woodlands, Conroe, Texas
  - Houston Methodist Cypress Hospital, Cypress, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - Houston Methodist West Hospital, Houston, Texas
  - MD Anderson League City, League City, Texas
  - Houston Methodist Saint John Hospital, Nassau Bay, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Westchester Emergency Center, Midlothian, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Richmond Community Hospital, Richmond, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Sheboygan Physicians Group, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
- Puerto Rico (4):
  - Doctors Cancer Center, Manatí
  - Centro Comprensivo de Cancer de UPR, San Juan
  - PROncology, San Juan
  - San Juan City Hospital, San Juan

IPD SHARING:
Plan to Share IPD: Undecided